CLINICAL TRIAL: NCT01551212
Title: A 12-month, Multi-center, Open-label, Randomized, Controlled Study to Evaluate Efficacy/Safety and Evolution of Renal Function of Everolimus in Co-exposure With Tacrolimus in de Novo Liver Transplant Recipients
Brief Title: Efficacy of Everolimus in Combination With Tacrolimus in Liver Transplant Recipients
Acronym: HEPHAISTOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001HDE13; 2011-003118-17 (EudraCT Number)
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation; Everolimus; Tacrolimus; Renal function
MeSH Terms: interventions — Everolimus; Tacrolimus; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVR/TAC (Experimental): Tacrolimus minimization arm. Everolimus (C0-h: 3-8 ng/mL) + tacrolimus (C0-h: < 5 ng/mL)
  Interventions: Drug: Everolimus; Drug: Tacrolimus; Drug: Corticosteroids
- TAC (Active Comparator): Tacrolimus (C0-h: 6-10 ng/ml)
  Interventions: Drug: Tacrolimus; Drug: Corticosteroids

INTERVENTIONS:
Drug: Everolimus — tablet containing 0.25mg, 0.5mg, 0.75mg or 1.0mg
  Other Names: RAD001 / Certican
  Arms: EVR/TAC
Drug: Tacrolimus — capsule containing 0.5, 1.0, or 5.0mg
  Other Names: Tacrolimus Hexal
Drug: Corticosteroids — For patients in all groups, corticosteroids were initiated at or prior to the time of transplantation according to local practice. Corticosteroids may have been used for the duration of the study according to the investigator's discretion, but may not have been eliminated sooner than 6 months post-transplantation.

SUMMARY:
This trial evaluated the efficacy and safety of Everolimus in combination with tacrolimus versus a standard immunosuppressive regimen concerning kidney function in liver transplant recipients.

ELIGIBILITY:
Inclusion criteria:

Male or female recipients of a full-size liver allograft, aged 18 to 65 years.

Exclusion criteria:

Patients with thrombocytopenia (platelets <50,000/mm³), with an absolute neutrophil count of <1,000/mm³ or leucopenia (leucocytes <2000/mm³), with anemia with Hb < 6g/dl at time of randomization

Patients with uncontrolled hypercholesterolemia (>350mg/dL; >9mmol/L) or hypertriglyceridemia (>750 mg/dL; >8.5 mmol/L) at time of randomization

History of malignancy of any organ system within the past 5 years whether or not there is evidence of local recurrence or metastases, other than non-metastatic basal or squamous cell carcinoma of the skin or HCC

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2012-05-24 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Germany (15):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Tübingen

REFERENCES:
- [Derived] Nashan B, Schemmer P, Braun F, Schlitt HJ, Pascher A, Klein CG, Neumann UP, Kroeger I, Wimmer P; Hephaistos Study Group. Early Everolimus-Facilitated Reduced Tacrolimus in Liver Transplantation: Results From the Randomized HEPHAISTOS Trial. Liver Transpl. 2022 Jun;28(6):998-1010. doi: 10.1002/lt.26298. Epub 2021 Oct 12. PMID 34525259
- [Derived] Nashan B, Schemmer P, Braun F, Dworak M, Wimmer P, Schlitt H. Evaluating the efficacy, safety and evolution of renal function with early initiation of everolimus-facilitated tacrolimus reduction in de novo liver transplant recipients: Study protocol for a randomized controlled trial. Trials. 2015 Mar 26;16:118. doi: 10.1186/s13063-015-0626-0. PMID 25873064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 642 patients were screened for study eligibility at 15 study centers in Germany. 339 patients were randomized out of which 333 received study treatment and were included in the analyses.
Pre-assignment Details: Patients were screened for eligibility prior to liver transplantation (LTx). The study treatment started after a run-in period that ended on the day of randomization, scheduled at Day 7-21 post-LTx. Patients may have been initiated on an optional induction therapy, MMF, TAC at investigators' discretion.
Groups:
- Everolimus/Tacrolimus: Tacrolimus minimization arm. Everolimus (C0-h: 3-8 ng/mL) + tacrolimus (C0-h: < 5 ng/mL)
- Tacrolimus: Tacrolimus (C0-h: 6-10 ng/ml)
Period: Overall Study
Arm/Group | Everolimus/Tacrolimus | Tacrolimus
Started (Randomized) | 171 | 168
Full Anylsis Set (FAS) (Randomized and received at least 1 dose of study drug) | 169 | 164
Safety Set (Received at least 1 dose of study drug and had a post-baseline safety assessment) | 169 | 164
Per Protocol Set (PP) (In FAS without a major protocol deviation) | 110 | 101
Completed | 166 | 148
Not Completed | 5 | 20
Not completed — Graft loss/Retransplantation | 0 | 1
Not completed — Administrative problems | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 7
Not completed — Death | 2 | 4
Not completed — Never Received Study Treatment | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus/Tacrolimus | Tacrolimus | Total
Number analyzed (Participants) | 169 | 164 | 333
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Full Analysis Set (FAS)
  Years | 53.68 (9.38) | 53.46 (9.64) | 53.57 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 79
  Male | 133 | 121 | 254
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Full Analysis Set (FAS)
  Participants
    Caucasian | 168 | 157 | 325
    Black | 1 | 1 | 2
    Asian | 0 | 3 | 3
    Other | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Estimated Glomerular Filtration Rate (GFR)
Description: The estmated GFR was calculated using MDRD-4 formula (Modification of Diet in Renal Disease Study Group).
Time Frame: month 12
Population: FAS (Full Analysis Set - All Randomized AND Treated Patients) with LOCF (last observation carried forward)
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Everolimus/Tacrolimus | Tacrolimus
Number analyzed (Participants) | 169 | 164
mL/min | 73.46 (25.57) | 71.95 (27.17)
Statistical Analysis 1: Comparison: Everolimus/Tacrolimus vs Tacrolimus; Test type: Superiority; p = 0.097, ANCOVA; factors: treatment, center, HCV-Class (positive, negative) and lab MELD (≤ 30 vs > 30) covariate: baseline value; Mean Difference (Final Values) = 4.09, 95% CI 2-sided [-0.74 to 8.91]

2. Secondary Outcome: Estimated GFR - PP Set
Description: This was a sensitivity analysis for the primary outcome measure based on the per-protocol set of patients.
Time Frame: month 12
Population: Per Protocol Set (PP)
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Everolimus/Tacrolimus | Tacrolimus
Number analyzed (Participants) | 110 | 101
mL/min | 74.83 (25.19) | 70.65 (24.91)
Statistical Analysis 1: Comparison: Everolimus/Tacrolimus vs Tacrolimus; Test type: Superiority; p = 0.0085, ANCOVA; factors: treatment, center, HCV-Class (positive, negative) and lab MELD (≤ 30 vs > 30) covariate: baseline value; Mean Difference (Final Values) = 7.99, 95% CI 2-sided [2.06 to 13.92]

3. Secondary Outcome: Percentage of Participants With Treated Biopsy Proven Acute Rejection (BPAR), Graft Loss or Death
Description: Percentage of Participants with Treated Biopsy Proven Acute Rejection (BPAR), Graft Loss or Death at Month 12
Time Frame: 12 months
Population: FAS
Measure: Number; unit: Percent of Patients
Arm/Group | Everolimus/Tacrolimus | Tacrolimus
Number analyzed (Participants) | 169 | 164
Percent of Patients | 9.5 | 7.9
Statistical Analysis 1: Comparison: Everolimus/Tacrolimus vs Tacrolimus; Test type: Superiority; p = 0.699, Fisher Exact

4. Secondary Outcome: Number of Participants With HCV
Description: Number of Participants with HCV (hepatitis C virus) assessed as treatment emergent adverse events of special interest
Time Frame: 12 months
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus/Tacrolimus | Tacrolimus
Number analyzed (Participants) | 169 | 164
Participants | 6 | 12

5. Secondary Outcome: Incidence of HCV Related Fibrosis
Description: Incidence of hepatitis C virus (HCV) related fibrosis assessed as treatment emergent adverse events of special interest
Time Frame: 12 months
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus/Tacrolimus | Tacrolimus
Number analyzed (Participants) | 169 | 164
Participants | 1 | 0

6. Secondary Outcome: Incidence of de Novo HCC Malignancies
Description: Incidence of de novo Hepatocellular Carcinoma (HCC) malignancies assessed as treatment emergent adverse events of special interest
Time Frame: 12 months
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus/Tacrolimus | Tacrolimus
Number analyzed (Participants) | 169 | 164
Participants | 0 | 2

7. Secondary Outcome: Incidence and Severity of CMV Viral Infections.
Description: Incidence and severity of cytomegalovirus (CMV) viral infections assessed as treatment emergent adverse events of special interest.
Time Frame: 12 months
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus/Tacrolimus | Tacrolimus
Number analyzed (Participants) | 169 | 164
Participants
  No CMV viral infection | 136 | 129
  Asymptomatic | 0 | 5
  Mild | 16 | 20
  Moderate | 13 | 9
  Severe | 4 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 12 months
Arm/Group | Everolimus/Tacrolimus | Tacrolimus
All-Cause Mortality (participants affected / at risk) | 3/169 | 4/164
Serious Adverse Events (participants affected / at risk) | 111/169 | 101/164
Other Adverse Events (participants affected / at risk) | 164/169 | 153/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus/Tacrolimus (N=169) | Tacrolimus (N=164)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 1
BONE MARROW TOXICITY (Blood and lymphatic system disorders) | 1 | 0
EVANS SYNDROME (Blood and lymphatic system disorders) | 0 | 1
HYPOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 3 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 3
TACHYCARDIA (Cardiac disorders) | 0 | 1
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
GOITRE (Endocrine disorders) | 1 | 0
TOXIC NODULAR GOITRE (Endocrine disorders) | 1 | 0
MYDRIASIS (Eye disorders) | 1 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 3 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 0
APHTHOUS ULCER (Gastrointestinal disorders) | 2 | 0
ASCITES (Gastrointestinal disorders) | 5 | 5
COLITIS (Gastrointestinal disorders) | 1 | 1
DENTAL CARIES (Gastrointestinal disorders) | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 5 | 4
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 1
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL ANGIODYSPLASIA HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 1 | 1
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 | 0
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 1
INTESTINAL INFARCTION (Gastrointestinal disorders) | 0 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
INTRA-ABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1 | 1
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 0 | 1
MESENTERIC VENOUS OCCLUSION (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 1
PANCREATITIS (Gastrointestinal disorders) | 2 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1
SUBILEUS (Gastrointestinal disorders) | 1 | 0
SWOLLEN TONGUE (Gastrointestinal disorders) | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 | 1
VOMITING (Gastrointestinal disorders) | 4 | 2
CHILLS (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 1
IMPAIRED HEALING (General disorders) | 1 | 3
INCARCERATED HERNIA (General disorders) | 1 | 0
MALAISE (General disorders) | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 1 | 0
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 2
PYREXIA (General disorders) | 4 | 2
SURGICAL FAILURE (General disorders) | 0 | 1
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1
BILE DUCT STENOSIS (Hepatobiliary disorders) | 5 | 6
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 1
BILIARY ISCHAEMIA (Hepatobiliary disorders) | 5 | 4
BILIARY TRACT DISORDER (Hepatobiliary disorders) | 0 | 1
BILOMA (Hepatobiliary disorders) | 2 | 2
CHOLANGITIS (Hepatobiliary disorders) | 13 | 7
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
CHOLESTASIS (Hepatobiliary disorders) | 1 | 4
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 | 1
HEPATIC ARTERY ANEURYSM (Hepatobiliary disorders) | 1 | 1
HEPATIC ARTERY STENOSIS (Hepatobiliary disorders) | 0 | 1
HEPATIC ARTERY THROMBOSIS (Hepatobiliary disorders) | 0 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 | 1
HEPATIC HAEMATOMA (Hepatobiliary disorders) | 1 | 0
HEPATIC HAEMORRHAGE (Hepatobiliary disorders) | 1 | 0
HEPATIC INFARCTION (Hepatobiliary disorders) | 1 | 0
HEPATIC ISCHAEMIA (Hepatobiliary disorders) | 0 | 1
HEPATIC LESION (Hepatobiliary disorders) | 0 | 1
HEPATIC NECROSIS (Hepatobiliary disorders) | 1 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 | 0
HEPATITIS TOXIC (Hepatobiliary disorders) | 0 | 1
HEPATOTOXICITY (Hepatobiliary disorders) | 0 | 1
LIVER DISORDER (Hepatobiliary disorders) | 1 | 0
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 1 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 | 2
VANISHING BILE DUCT SYNDROME (Hepatobiliary disorders) | 0 | 1
LIVER TRANSPLANT REJECTION (Immune system disorders) | 12 | 9
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 1
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 | 1
ABSCESS JAW (Infections and infestations) | 1 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 1
APPENDICITIS (Infections and infestations) | 1 | 0
ATYPICAL PNEUMONIA (Infections and infestations) | 1 | 2
BACTERAEMIA (Infections and infestations) | 0 | 1
BACTERIAL INFECTION (Infections and infestations) | 1 | 0
BILIARY ABSCESS (Infections and infestations) | 0 | 1
BILIARY TRACT INFECTION (Infections and infestations) | 0 | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 0
CHOLANGITIS INFECTIVE (Infections and infestations) | 6 | 1
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 2 | 0
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 1 | 2
CYTOMEGALOVIRUS HEPATITIS (Infections and infestations) | 1 | 0
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 6 | 3
CYTOMEGALOVIRUS SYNDROME (Infections and infestations) | 1 | 0
CYTOMEGALOVIRUS VIRAEMIA (Infections and infestations) | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 1
EMPYEMA (Infections and infestations) | 0 | 1
ENTERITIS INFECTIOUS (Infections and infestations) | 1 | 0
ENTEROCOCCAL INFECTION (Infections and infestations) | 1 | 1
EPIDIDYMITIS (Infections and infestations) | 0 | 1
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 0 | 1
ESCHERICHIA INFECTION (Infections and infestations) | 1 | 0
FEBRILE INFECTION (Infections and infestations) | 0 | 1
FOLLICULITIS (Infections and infestations) | 1 | 1
FUNGAL INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 3 | 1
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 1 | 0
GASTROENTERITIS CRYPTOSPORIDIAL (Infections and infestations) | 0 | 1
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 0 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 1
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 0 | 1
HAEMATOMA INFECTION (Infections and infestations) | 2 | 3
HEPATITIS C (Infections and infestations) | 2 | 5
HERPES ZOSTER (Infections and infestations) | 0 | 2
HUMAN HERPESVIRUS 6 INFECTION (Infections and infestations) | 1 | 0
INFECTED SEROMA (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 4 | 3
LIVER ABSCESS (Infections and infestations) | 5 | 4
LOCALISED INFECTION (Infections and infestations) | 0 | 1
LUNG INFECTION (Infections and infestations) | 0 | 1
PARONYCHIA (Infections and infestations) | 1 | 0
PERITONITIS (Infections and infestations) | 1 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 2 | 1
PHARYNGEAL ABSCESS (Infections and infestations) | 0 | 1
PILONIDAL CYST (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 10 | 7
PSEUDOMONAS INFECTION (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
SCARLET FEVER (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 2 | 4
SEPTIC SHOCK (Infections and infestations) | 2 | 3
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
TRANSPLANT ABSCESS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 2 | 5
VARICELLA (Infections and infestations) | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0
WOUND INFECTION (Infections and infestations) | 3 | 0
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 | 0
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 3 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 1
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 1 | 1
BILIARY ANASTOMOSIS COMPLICATION (Injury, poisoning and procedural complications) | 8 | 13
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
COMPLICATIONS OF TRANSPLANTED LIVER (Injury, poisoning and procedural complications) | 1 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
GRAFT LOSS (Injury, poisoning and procedural complications) | 0 | 1
INCARCERATED INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 11 | 4
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 2 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL BILE LEAK (Injury, poisoning and procedural complications) | 1 | 3
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TRANSPLANT FAILURE (Injury, poisoning and procedural complications) | 0 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 | 1
WEANING FAILURE (Injury, poisoning and procedural complications) | 1 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 2
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 3 | 3
BLOOD POTASSIUM INCREASED (Investigations) | 2 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 5
CHEST X-RAY ABNORMAL (Investigations) | 0 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 | 1
GLUTAMATE DEHYDROGENASE INCREASED (Investigations) | 1 | 1
HAEMOGLOBIN DECREASED (Investigations) | 2 | 1
HEPATIC ARTERY FLOW DECREASED (Investigations) | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 6 | 7
LIVER FUNCTION TEST INCREASED (Investigations) | 3 | 0
TRANSAMINASES INCREASED (Investigations) | 2 | 6
TROPONIN INCREASED (Investigations) | 0 | 1
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 | 1
ACIDOSIS HYPERCHLORAEMIC (Metabolism and nutrition disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
DIABETIC COMPLICATION (Metabolism and nutrition disorders) | 1 | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 1 | 1
GOUT (Metabolism and nutrition disorders) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPERINSULINAEMIC HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 1
EPILEPSY (Nervous system disorders) | 1 | 1
HEMIPARESIS (Nervous system disorders) | 0 | 1
LACUNAR STROKE (Nervous system disorders) | 0 | 1
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 | 1
PARAPARESIS (Nervous system disorders) | 0 | 1
POLYNEUROPATHY (Nervous system disorders) | 0 | 1
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 1 | 0
SEIZURE (Nervous system disorders) | 2 | 0
SYNCOPE (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 1
TREMOR (Nervous system disorders) | 0 | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 1
DEVICE OCCLUSION (Product Issues) | 1 | 1
DISORIENTATION (Psychiatric disorders) | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 10 | 8
ALBUMINURIA (Renal and urinary disorders) | 1 | 0
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 | 1
IGA NEPHROPATHY (Renal and urinary disorders) | 0 | 1
OLIGURIA (Renal and urinary disorders) | 1 | 0
PRERENAL FAILURE (Renal and urinary disorders) | 0 | 1
PROTEINURIA (Renal and urinary disorders) | 2 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 2
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 2
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 | 5
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 | 0
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0
ANGIODYSPLASIA (Vascular disorders) | 1 | 0
ARTERY DISSECTION (Vascular disorders) | 0 | 1
DIABETIC VASCULAR DISORDER (Vascular disorders) | 1 | 0
HAEMATOMA (Vascular disorders) | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 1
INFERIOR VENA CAVA STENOSIS (Vascular disorders) | 1 | 0
INTERNAL HAEMORRHAGE (Vascular disorders) | 1 | 0
LYMPHATIC FISTULA (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 | 1
POOR PERIPHERAL CIRCULATION (Vascular disorders) | 0 | 1
THROMBOSIS (Vascular disorders) | 2 | 0
VENA CAVA THROMBOSIS (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus/Tacrolimus (N=169) | Tacrolimus (N=164)
ANAEMIA (Blood and lymphatic system disorders) | 22 | 20
LEUKOPENIA (Blood and lymphatic system disorders) | 45 | 12
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 25 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 23 | 17
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 15 | 11
APHTHOUS ULCER (Gastrointestinal disorders) | 11 | 0
ASCITES (Gastrointestinal disorders) | 20 | 13
CONSTIPATION (Gastrointestinal disorders) | 13 | 10
DIARRHOEA (Gastrointestinal disorders) | 43 | 39
NAUSEA (Gastrointestinal disorders) | 22 | 13
VOMITING (Gastrointestinal disorders) | 16 | 12
IMPAIRED HEALING (General disorders) | 24 | 10
OEDEMA PERIPHERAL (General disorders) | 38 | 15
PYREXIA (General disorders) | 20 | 9
CHOLANGITIS (Hepatobiliary disorders) | 9 | 2
HEPATIC CYST (Hepatobiliary disorders) | 10 | 3
HEPATIC STEATOSIS (Hepatobiliary disorders) | 12 | 8
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 24 | 28
URINARY TRACT INFECTION (Infections and infestations) | 30 | 24
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 41 | 29
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 35 | 10
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 5 | 9
BLOOD CREATININE INCREASED (Investigations) | 21 | 21
BODY TEMPERATURE INCREASED (Investigations) | 6 | 9
C-REACTIVE PROTEIN INCREASED (Investigations) | 18 | 9
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 10 | 12
HEPATIC ENZYME INCREASED (Investigations) | 9 | 13
TRANSAMINASES INCREASED (Investigations) | 9 | 8
DIABETES MELLITUS (Metabolism and nutrition disorders) | 11 | 8
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 30 | 9
HYPERKALAEMIA (Metabolism and nutrition disorders) | 13 | 17
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 15 | 2
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 18 | 8
HYPERURICAEMIA (Metabolism and nutrition disorders) | 10 | 8
HYPOKALAEMIA (Metabolism and nutrition disorders) | 11 | 8
IRON DEFICIENCY (Metabolism and nutrition disorders) | 11 | 5
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 11 | 10
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9 | 8
BACK PAIN (Musculoskeletal and connective tissue disorders) | 17 | 12
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 7 | 9
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 | 5
HEADACHE (Nervous system disorders) | 48 | 22
TREMOR (Nervous system disorders) | 25 | 23
DEPRESSION (Psychiatric disorders) | 4 | 10
INSOMNIA (Psychiatric disorders) | 1 | 9
PROTEINURIA (Renal and urinary disorders) | 26 | 12
RENAL FAILURE (Renal and urinary disorders) | 12 | 15
RENAL IMPAIRMENT (Renal and urinary disorders) | 7 | 15
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 | 8
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 | 7
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 20 | 12
ALOPECIA (Skin and subcutaneous tissue disorders) | 10 | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 16 | 10
HYPERTENSION (Vascular disorders) | 28 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-08-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT01551212/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT01551212/SAP_001.pdf